CLINICAL TRIAL: NCT05588804
Title: A Randomized Double-blind Placebo-controlled Comparative Multicenter Study of the Efficacy and Safety of Broncho-munal®, Capsules, 7 mg (Sandoz dd, Slovenia) in the Treatment of Patients With Acute Uncomplicated Respiratory Tract Infections
Brief Title: Study of the Efficacy and Safety of Broncho-munal®, Capsules, 7 mg for the Treatment of Acute Uncomplicated Respiratory Tract Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CT_003_BRO_CAP/SAN-0632
Record Dates: First submitted 2022-10-17; First posted 2022-10-20 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Acute Uncomplicated Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Broncho-munal® (Experimental): Participants will receive the study drug Broncho-munal®, capsules, 7 mg (Sandoz dd, Slovenia), 1 capsule per day in the morning on an empty stomach, 30 minutes before meals, for 10 consecutive days
  Interventions: Drug: Broncho-munal®
- Group 2: Placebo (Placebo Comparator): Participants will receive a placebo, 1 capsule per day in the morning on an empty stomach, 30 minutes before meals, for 10 consecutive days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Broncho-munal® — 1 capsule daily in the morning on an empty stomach, 30 minutes before meals, for 10 consecutive days
  Arms: Group 1: Broncho-munal®
Drug: Placebo — 1 capsule daily in the morning on an empty stomach, 30 minutes before meals, for 10 consecutive days
  Arms: Group 2: Placebo

SUMMARY:
The study will evaluate the efficacy and safety of Broncho-munal®, capsules, 7 mg (Sandoz dd, Slovenia) versus Placebo in the treatment of patients with acute uncomplicated respiratory tract infections.

DETAILED DESCRIPTION:
Patients who meet the inclusion criteria and do not meet the exclusion criteria will be randomized into 2 groups in a 1: 1 ratio.

Group 1 (n = 278) will receive the study drug Broncho-munal®, capsules, 7 mg (Sandoz dd, Slovenia),

Group 2 (n = 278) will receive a placebo

ELIGIBILITY:
Inclusion Criteria:

* Patient signing and dating of the Patient Information Sheet Informed Consent Form.
* Men and women between the ages of 18 and 60 inclusive at the time of signing the Patient Information Sheet Informed Consent Form.
* Symptoms of acute uncomplicated respiratory tract infection of mild to moderate severity:
* The presence of two or more symptoms of moderate severity or three or more symptoms of mild severity according to the WURSS-21 questionnaire
* The presence of two or more symptoms of moderate severity or three or more symptoms of mild severity according to the CCQ questionnaire
* Body temperature ≥ 37.50 ° C and ≤ 40.0 ° C since the onset of the disease.
* Duration of disease symptoms less than 36 hours prior to randomization.
* The patient's consent to use reliable contraceptive methods throughout the study and for 3 weeks after its completion. The following may take part in the study:

women who have a negative pregnancy test and are using the following contraception: barrier method (condom or occlusion cap (diaphragm or cervical / vaulted cap)) or dual barrier method of contraception (condom or occlusive cap (diaphragm or cervical / sperm cap (cid) plus foam / gel / film / cream / suppository)). The study may also include women who are unable to bear children.

(history: hysterectomy, tubal ligation, infertility, menopause for more than 1 year).

Or men with safe reproductive function using barrier contraception, as well as men with infertility or previous vasectomy history.

Exclusion Criteria:

* Aggravated history of allergies, including food allergies
* Intolerance to drugs, incl. hypersensitivity or idiosyncrasy to Broncho-munal® or its excipients and to any other product from the concomitant / standard treatment
* A positive result of the analysis performed by the PCR method for the presence of SARS-CoV-2 RNA at the screening stage.
* Positive result of the analysis performed by Rapid Influenza Diagnostic Test for the presence of the influenza virus at the screening stage.
* Clinically confirmed of the presence of a new coronavirus infection COVID-19 in accordance with the regulatory acts of the Ministry of Health of the Russian Federation for the prevention, diagnosis and treatment of a new coronavirus infection (COVID-19), (the version is current at the time of inclusion of patients).
* Any vaccination less than 30 days before screening.
* The presence of any symptom of a severe course of the disease (fever of 40 ° C and higher, pulse - more than 120 beats / min, SBP - less than 90 mm Hg, muffled heart sounds, NPV - more than 28 per minute, the presence of complications, impairment of consciousness, seizures).
* Other infectious diseases less than 14 days before the screening visit, including those requiring local and / or systemic antibiotic therapy (cystitis, pyelonephritis, endocarditis, etc.)
* Chronic lung diseases (such as cystic fibrosis, pulmonary emphysema, tracheobchonchial dyskinesia, chronic obstructive pulmonary disease (COPD), bronchiectasis, etc.) in the acute stage.
* Bronchial asthma and chronic bronchitis in history.
* Pulmonary tuberculosis (active or inactive form).
* The use of drugs with immunomodulatory (including Broncho-munal) and / or immunostimulating and / or immunosuppressive effects, less than 1 month before screening.
* The need to use drugs from the list of prohibited therapy.
* Peptic ulcer of the stomach and duodenum or other erosive and ulcerative lesions of the gastrointestinal tract in the acute stage.
* Syndrome of malabsorption or other clinically significant disease of the gastrointestinal tract (uncorrected vomiting, diarrhea, ulcerative colitis, and others).
* Deficiency of the enzyme glucose-6-phosphate dehydrogenase.
* Dehydration, hypovolemia, anorexia, bulimia and cachexia (insufficient supply of glutathione in the liver) according to the anamnesis at the time of screening.
* Autoimmune diseases, according to anamnesis (systemic lupus erythematosus, rheumatoid arthritis, etc.).
* Uncontrolled diabetes mellitus.
* Syndrome of renal or hepatic insufficiency, confirmed by physical examination data.
* Positive result of any of the following tests: blood test for Hep. B, Hep.C, HIV and/or syphillis.
* Chronic heart failure III - IV functional class according to the functional classification of the New York Heart Association (NYHA), including unstable progressive angina pectoris IV functional class, uncontrolled arterial hypertension, severe arterial hypotension.
* A history of malignant neoplasms.
* Alcohol or drug addiction, history of mental illness.
* Smoking more than 20 cigarettes a day.
* Severe, decompensated or unstable somatic diseases (any diseases or conditions that threaten the patient's life or worsen the patient's prognosis, as well as make it impossible for him to participate in a clinical trial).
* Major surgery, 3 months before screening (associated with a risk to the patient's life).
* Patient's unwillingness or inability to comply with Protocol procedures (in the opinion of the investigator).
* Taking other medications that, in the Investigator's opinion, may affect the course and results of the clinical trial.
* Pregnancy or breastfeeding period.
* Participation in other clinical trials at the screening visit or for 30 days before the screening visit.
* Other conditions that, in the Investigator's opinion prevent the patient from being included in the research.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 556 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2022-12-18 (Actual); Study Completion 2022-12-18 (Actual)

PRIMARY OUTCOMES:
AUC value of the change in the symptom severity according to the WURSS-21 questionnaire | by 3, 5, 7 and 10 days after the start of therapy
  Dynamics of symptoms severity according to the WURSS-21 is assessed using the Area under the curve (AUC) for the score for 3, 5, 7 and 10 days of the treatment.
  WURSS-21 consists of 21 items (2 questions and 2 domains. Symptoms domain consists of 10 items: Runny nose, Plugged nose, Sneezing, Sore throat, Scratchy throat, Cough, Hoarseness, Head congestion, Chest congestion, Feeling tired. Ability domain consists of 9 items: Think clearly, Sleep well, Breathe easily, Walk, climb stairs, exercise, Accomplish daily activities, Work outside the home, Work inside the home, Interact with others, Live your personal life. The first 20 items are scored according to the 8-point scale (from 0 to 7). The last item is scored according to the 7-point scale: (from 0 to 6). Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Change in symptom severity index according to the WURSS-21 questionnaire | by 3, 5, 7 and 10 days after the start of therapy
  WURSS-21 consists of 21 items (2 questions and 2 domains. Symptoms domain consists of 10 items: Runny nose, Plugged nose, Sneezing, Sore throat, Scratchy throat, Cough, Hoarseness, Head congestion, Chest congestion, Feeling tired. Ability domain consists of 9 items: Think clearly, Sleep well, Breathe easily, Walk, climb stairs, exercise, Accomplish daily activities, Work outside the home, Work inside the home, Interact with others, Live your personal life. The first 20 items are scored according to the 8-point scale (from 0 to 7). The last item is scored according to the 7-point scale: (from 0 to 6). Higher scores mean a worse outcome.
Change in symptom severity index on the CCQ scale | by 3, 5, 7 and 10 days after the start of therapy
  General symptoms (fever, chills, muscle pain), nasal symptoms (nasal discharge, sneezing, watery eyes), throat (sore throat) and chest symptoms (cough, chest pain) are assessed in points from 0 to 3. Assessment will be conducted by the Investigating Physician during visits to the Research Center. A ´probable' viral infection is where there are moderate symptoms noted in at least 2 of the above 4 categories or mild symptoms noted in 3 or more categories. A ´possible´ viral infection is where mild symptoms are noted in one category plus a cough. Scoring: none=0, mild=1, moderate=2 and severe=3. Total score equals the sum of all scores.
Time (in days) until the symptoms of the disease disappear according to the WURSS-21 scale | by 3, 5, 7 and 10 days after the start of therapy
  WURSS-21 consists of 21 items (2 questions and 2 domains. Symptoms domain consists of 10 items: Runny nose, Plugged nose, Sneezing, Sore throat, Scratchy throat, Cough, Hoarseness, Head congestion, Chest congestion, Feeling tired. Ability domain consists of 9 items: Think clearly, Sleep well, Breathe easily, Walk, climb stairs, exercise, Accomplish daily activities, Work outside the home, Work inside the home, Interact with others, Live your personal life. The first 20 items are scored according to the 8-point scale (from 0 to 7). The last item is scored according to the 7-point scale: (from 0 to 6). Higher scores mean a worse outcome.
Time (in days) until symptoms disappear on the CCQ scale | by 3, 5, 7 and 10 days after the start of therapy
  General symptoms (fever, chills, muscle pain), nasal symptoms (nasal discharge, sneezing, watery eyes), throat (sore throat) and chest symptoms (cough, chest pain) are assessed in points from 0 to 3. Assessment will be conducted by the Investigating Physician during visits to the Research Center. A ´probable' viral infection is where there are moderate symptoms noted in at least 2 of the above 4 categories or mild symptoms noted in 3 or more categories. A ´possible´ viral infection is where mild symptoms are noted in one category plus a cough. Scoring: none=0, mild=1, moderate=2 and severe=3. Total score equals the sum of all scores.
Total score on the WURSS-21 scale | by 3, 5, 7 and 10 days after the start of therapy
  WURSS-21 consists of 21 items (2 questions and 2 domains. Symptoms domain consists of 10 items: Runny nose, Plugged nose, Sneezing, Sore throat, Scratchy throat, Cough, Hoarseness, Head congestion, Chest congestion, Feeling tired. Ability domain consists of 9 items: Think clearly, Sleep well, Breathe easily, Walk, climb stairs, exercise, Accomplish daily activities, Work outside the home, Work inside the home, Interact with others, Live your personal life. The first 20 items are scored according to the 8-point scale (from 0 to 7). The last item is scored according to the 7-point scale: (from 0 to 6). Higher scores mean a worse outcome.
Total score on the CCQ scale | by 3, 5, 7 and 10 days after the start of therapy
  General symptoms (fever, chills, muscle pain), nasal symptoms (nasal discharge, sneezing, watery eyes), throat (sore throat) and chest symptoms (cough, chest pain) are assessed in points from 0 to 3. Assessment will be conducted by the Investigating Physician during visits to the Research Center. A ´probable' viral infection is where there are moderate symptoms noted in at least 2 of the above 4 categories or mild symptoms noted in 3 or more categories. A ´possible´ viral infection is where mild symptoms are noted in one category plus a cough. Scoring: none=0, mild=1, moderate=2 and severe=3. Total score equals the sum of all scores.
Number of patients with symptoms and daily activity of varying severity on the WURSS-21 scale | by 3, 5, 7 and 10 days after the start of therapy
  WURSS-21 consists of 21 items (2 questions and 2 domains. Symptoms domain consists of 10 items: Runny nose, Plugged nose, Sneezing, Sore throat, Scratchy throat, Cough, Hoarseness, Head congestion, Chest congestion, Feeling tired. Ability domain consists of 9 items: Think clearly, Sleep well, Breathe easily, Walk, climb stairs, exercise, Accomplish daily activities, Work outside the home, Work inside the home, Interact with others, Live your personal life. The first 20 items are scored according to the 8-point scale (from 0 to 7). The last item is scored according to the 7-point scale: (from 0 to 6). Higher scores mean a worse outcome.
Number of patients with symptoms of varying severity on the CCQ scale | by 3, 5, 7 and 10 days after the start of therapy
  General symptoms (fever, chills, muscle pain), nasal symptoms (nasal discharge, sneezing, watery eyes), throat (sore throat) and chest symptoms (cough, chest pain) are assessed in points from 0 to 3. Assessment will be conducted by the Investigating Physician during visits to the Research Center. A ´probable' viral infection is where there are moderate symptoms noted in at least 2 of the above 4 categories or mild symptoms noted in 3 or more categories. A ´possible´ viral infection is where mild symptoms are noted in one category plus a cough. Scoring: none=0, mild=1, moderate=2 and severe=3. Total score equals the sum of all scores.
Number of patients with complete disappearance of symptoms according to the WURSS-21 questionnaire for each day of therapy | by 3, 5, 7 and 10 days after the start of therapy
  WURSS-21 consists of 21 items (2 questions and 2 domains. Symptoms domain consists of 10 items: Runny nose, Plugged nose, Sneezing, Sore throat, Scratchy throat, Cough, Hoarseness, Head congestion, Chest congestion, Feeling tired. Ability domain consists of 9 items: Think clearly, Sleep well, Breathe easily, Walk, climb stairs, exercise, Accomplish daily activities, Work outside the home, Work inside the home, Interact with others, Live your personal life. The first 20 items are scored according to the 8-point scale (from 0 to 7). The last item is scored according to the 7-point scale: (from 0 to 6). Higher scores mean a worse outcome.
Number of patients with complete disappearance of symptoms on the CCQ scale for each day of therapy | by 3, 5, 7 and 10 days after the start of therapy
  General symptoms (fever, chills, muscle pain), nasal symptoms (nasal discharge, sneezing, watery eyes), throat (sore throat) and chest symptoms (cough, chest pain) are assessed in points from 0 to 3. Assessment will be conducted by the Investigating Physician during visits to the Research Center. A ´probable' viral infection is where there are moderate symptoms noted in at least 2 of the above 4 categories or mild symptoms noted in 3 or more categories. A ´possible´ viral infection is where mild symptoms are noted in one category plus a cough. Scoring: none=0, mild=1, moderate=2 and severe=3. Total score equals the sum of all scores.
Number of patients with body temperature <37°C from the moment the temperature drops to completion of therapy for each day of therapy | by 3, 5, 7 and 10 days after the start of therapy
  Number of patients with body temperature <37°C from the moment the temperature drops to completion of therapy for each day of therapy will be reported.
Number of patients with the need for systemic antibiotic therapy | by 3, 5, 7 and 10 days after the start of therapy
  Number of patients requiring local and / or systemic antibiotic therapy (cystitis, pyelonephritis, endocarditis, etc.) will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Sandoz, Study Director — Sandoz
Locations (3):
- Russia (3):
  - Sandoz Investigative Site, Moscow
  - Sandoz Investigative Site, Nizhny Novgorod
  - Sandoz Investigative Site, Saint Petersburg

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.